CLINICAL TRIAL: NCT02266628
Title: A Phase II Randomized, Observer-Blind, Placebo- Controlled Study to Evaluate the Immunogenicity and Safety of Respiratory Syncytial Virus (RSV) F Vaccine in Healthy Elderly Subjects and to Estimate the Incidence Rate of Medically-attended RSV Disease in Vaccine and Placebo Recipients
Brief Title: Placebo- Controlled Study to Evaluate the Safety and Immunogenicity of the RSV-F Vaccine in Elderly Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RSV-E-201
Record Dates: First submitted 2014-10-13; First posted 2014-10-17 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (Experimental): RSV-F vaccine (0.5mL Injection)
  Interventions: Biological: RSV-F Vaccine
- Treatment Group B (Placebo Comparator): Saline Placebo (0.5mL Injection)
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: RSV-F Vaccine
  Arms: Treatment Group A
Biological: Saline Placebo
  Arms: Treatment Group B

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the RSV- F Vaccine in elderly subjects, as well as rate the incidence of medically- attended RSV disease in vaccine and placebo recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥60 years of age who are ambulatory and live in the community or in residential facilities which provide minimal assistance, such that the subject is primarily responsible for self-care and activities of daily living. Subjects may have one or more chronic medical diagnoses, but should be clinically stable as assessed by:

   * Absence of changes in medical therapy within one month due to treatment failure or toxicity,
   * Absence of medical events qualifying as serious adverse events (SAEs) within two months, and
   * Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the investigator.
2. Willing and able (on both a physical and cognitive basis) to give informed consent prior to study enrollment.
3. Able to comply with study requirements; including access to transportation for study visits.
4. Access to inbound and outbound telephone communication with caregivers and study staff.

Exclusion Criteria:

1. Participation in research involving investigational product (drug / biologic / device) within 45 days before the planned date of the Day 0 vaccination.
2. History of a serious reaction to any prior vaccination, or Guillain-Barré syndrome within 6 weeks of any prior influenza immunization.
3. Received any vaccine other than an inactivated influenza vaccine in the 4 weeks preceding the study vaccination; or any RSV vaccine at any time.
4. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
5. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
6. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
7. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥38.0°C on the planned day of vaccine administration).
8. Known disturbance of coagulation.
9. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
10. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic, cognitive, or psychiatric conditions deemed likely to impair the quality of study compliance or safety reporting).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1599 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Immunogenicity as assessed by serum IgG antibody titers specific for the F-Protein antigen | Day 0 to Day 364
  Serum IgG antibody concentrations as ELISA units (EUs) specific for the F protein antigen. Derived/ calculated endpoints based on these data will include:
  * Geometric mean concentrations as EU (GMEU)
  * Geometric mean ratio (GMR)
  * Geometric mean fold-rise( GMFR)
  * Seroresponse rate (SRR)
Number and percentage of subjects with respiratory illness associated with RSV | Day 0 to Day 364
  Defined by any one of rhinorrhea, nasal congestion, pharyngitis, cough, wheezing (or increase in baseline wheezing), sputum production (or increase in the change in nature of baseline sputum production), or new (or worsening) shortness of breath; plus RT-PRC-confirmed RSV infection documented within three days of symptom onset.
Numbers and percentages of subjects with solicited local and systemic AEs. | Day 0 to Day 364
  Solicited local and systemic AEs over the seven days post-injection; and all adverse events, solicited and unsolicited, including adverse changes in clinical laboratory parameters over 56 days post injection. In addition, MAEs, SAEs, and SNMCs will be collected for one year.

SECONDARY OUTCOMES:
Palivizumab competitive antibody responses based on antibody titers in competitive ELISA. | Day 0 to Day 182
  Summarized by geometric mean titer (GMT), GMR. GMFR, and SRR; as well as seroconversion rate (SCR).
Neutralizing antibody titer to at least one prototypical RSV/A and one RSV/B virus strain. | Day 0 to Day 182
  Analyzed by GMT,GMR, SCR, and SRR. Neutralizing antibody assays, because of their time intensive nature, will be performed at a selected subset of time-points.
Hemagglutination-inhibiting (HAI) antibody titers specific for the viruses in the 2014-15 vaccine at Day 28. | Day 0 to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (10):
- United States (10):
  - Nothern California Clinical Research, Redding, California
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Rapid Medical Research, Cleveland, Ohio
  - Clinical Research Associates, Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Lisa Jackson, Seattle, Washington
  - Marshfield Clinical Research Foundation, Wausau, Wisconsin